CLINICAL TRIAL: NCT06971185
Title: Treatment Patterns and Effectiveness of Luspatercept in the Real World
Brief Title: A Study to Evaluate Treatment Patterns and Effectiveness of Luspatercept
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1124
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Myelodysplastic syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept; Hematinics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Participants treated with first-line (1L) luspatercept treatment
  Interventions: Drug: Luspatercept
- Cohort 2: Participants treated with first-line (1L) erythropoiesis stimulating agents
  Interventions: Drug: Erythropoiesis-stimulating agent (ESA)
- Cohort 3: Participants treated with second-line (2L) luspatercept treatment
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — As per product label
  Groups: Cohort 1; Cohort 3
Drug: Erythropoiesis-stimulating agent (ESA) — As per product label
  Groups: Cohort 2

SUMMARY:
The purpose of this study is to understand the treatment patterns and clinical outcomes of myelodysplastic syndromes patients treated with luspatercept or erythropoiesis-stimulating agents

ELIGIBILITY:
Inclusion Criteria:

* Included in the Flatiron Health Broad Research Network, with 2 or more visits after January 1, 2011
* Has evidence of diagnosis with myelodysplastic syndromes (MDS) after Jan 1, 2020, as identified by a natural language processing (NLP)-based machine-learning (ML) model
* Has evidence of diagnosis with MDS as identified via structured International Classification of Diseases (ICD) codes:

  * International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM): D46.x
  * International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM): 238.7x
* Age ≥ 18 years at MDS diagnosis
* Has either ring sideroblasts positive or negative status, as confirmed by bone marrow aspirate lab results or clinician notes
* Has at least one confirmed structured activity more than 8 weeks prior to the index date

Cohort specific inclusion criteria:

First-line (1L) luspatercept cohort

* Has evidence of receipt of luspatercept as identified via structured data as evidenced by non-cancelled Medication Order or Medication Administration and confirmed via unstructured data
* Has evidence of treatment with luspatercept for at least 12 weeks as evidenced by non-cancelled Medication Orders or Medication Administrations

  1L erythropoiesis stimulating agents (ESA) cohort:
* Has evidence of receipt of any ESA (i.e., epoetin alfa, darbepoetin alfa, epoetin beta, epoetin alfa-epbx, epoetin zeta, or epoetin beta-methoxy polyethylene glycol) for at least 12 weeks as evidenced by non-cancelled Medication Orders or Medication Administrations
* Note: this criterion is included to maximize alignment between the 1L ESA cohort and the 1L luspatercept cohort and minimize bias induced by the dosage requirement in the 1L luspatercept cohort

Second-lin (2L) luspatercept cohort:

* Has evidence of receipt of luspatercept as identified via structured data as evidenced by non-cancelled Medication Order or Medication Administration and confirmed via unstructured data
* Has evidence of receipt of at least 1 ESA as evidenced by a non-cancelled medication order or medication administration prior to the date of initial luspatercept receipt
* Has evidence of treatment with luspatercept for at least 12 weeks as evidenced by non-cancelled Medication Orders or Medication Administrations

Exclusion Criteria:

* Lacking relevant unstructured documents in the Flatiron database for review by the abstraction team
* Have been exposed to any of the following MDS-related therapy prior to luspatercept initiation in the 1L and 2L settings or ESA initiation in the 1L setting: lenalidomide, azacitidine, decitabine, cedazuridine, eltrombopag, cytarabine, daunorubicin, idarubicin, filgrastim, pegfilgrastim, lipefilgrastim, sargramostim, venetoclax, or has evidence of a stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients identified from the Flatiron Health electronic health record database between January 1, 2011 and August 31, 2024 that have been diagnosed with myelodysplastic syndromes receiving either (a) first-line (1L) luspatercept, (b) 1L erythropoiesis stimulating agents, or (c) second-line luspatercept treatment.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Luspatercept dose at treatment initiation | Baseline
  Cohort 1 and 3 only
Luspatercept dose at treatment discontinuation | Up to 50 months
  Cohort 1 and 3 only
Luspatercept dose change or escalation or reduction | Up to 50 months
  Cohort 1 and 3 only
Time from luspatercept initiation to the first occurrence of dose escalation | Up to 50 months
  Cohort 1 and 3 only
Proportion of participants that discontinued treatment | Up to 50 months
Time from treatment initiation to treatment discontinuation | Up to 50 months
Time from luspatercept/erythropoiesis stimulating agents treatment initiation to initiation of a new treatment for myelodysplastic syndromes | Up to 50 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol Myers Squibb, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts